CLINICAL TRIAL: NCT00185640
Title: Allogeneic Hematopoietic Cell Transplantation Using a Non-Myeloablative Preparative Regimen of Total Lymphoid Irradiation and Anti-Thymocyte Globulin for Older Patients With Hematologic Malignancies
Brief Title: Allogeneic Transplantation Using Total Lymphoid Irradiation (TLI) and Anti-Thymocyte Globulin (ATG) for Older Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Lowsky, Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-11960; 78998 (Other: Stanford University Alternate IRB Approval Number); BMT153 (Other: OnCore); NCT00186615 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Blood Cancer; Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia | interventions — Cyclosporine; Antilymphocyte Serum; thymoglobulin; Mycophenolic Acid; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-myeloablative transplantation (Experimental): Pre-transplant total lymphoid irradiation (TLI) and anti-thymocyte globulin (ATG) infusion with Day 0 allogeneic hematopoietic cell transplant (HCT), followed by post-transplant immunosuppression by cyclosporine and mycophenolate mofetil.
  Interventions: Drug: Cyclosporine; Drug: Anti-thymocyte globulin (ATG); Drug: Mycophenolate mofetil (MMF); Drug: Filgrastim; Radiation: Total Lymphoid Irradiation (TLI)

INTERVENTIONS:
Drug: Cyclosporine — Starting day -3 at a dose of 5 mg/kg orally twice daily with a target trough level of 350 to 450 ng/mL
  Other Names: Cyclosporin; Cyclosporin A
Drug: Anti-thymocyte globulin (ATG) — 1.5 mg/kg for total dose of 7.5mg/kg, IV starting on day -11 to day -7 before HCT
  Other Names: Thymoglobulin
Drug: Mycophenolate mofetil (MMF) — Begins on day 0 after HCT at a dose of 15 mg/kg. Transplant recipients who received related donor grafts received MMF twice daily and those who received unrelated donor grafts received MMF 3 times daily.
  Other Names: CellCept
Drug: Filgrastim — * Donors mobilized with 16 µg/kg/day filgrastim.
  * As needed, myelosuppression in transplant recipients will be managed with subcutaneous filgrastim 5 µg/kg/day
  Other Names: Neupogen; Granulocyte-colony stimulating factor (G-CSF; GCSF); colony-stimulating factor 3 (CSF-3)
Radiation: Total Lymphoid Irradiation (TLI) — 0.8 Gy/day from day -11 to day -7 (inclusive) from day -4 to day -2 (inclusive) with 2 additional fractions of 0.8 Gy delivered on day -1 for total dose of 8 Gy.

SUMMARY:
To measure how frequently and to what degree a complication of transplant cell acute graft versus host disease (GvHD) occurs.

DETAILED DESCRIPTION:
This study evaluated whether TLI-ATG conditioning followed by allogeneic hematpoietic cell transplant (HCT), which has provided excellent overall survival for patients with relapsed lymphoma after failed autologous HCT, provides a similar benefit in the setting of elderly patients with hematologic malignancies.

ELIGIBILITY:
INCLUSION CRITERIA:

* Any patient with one of the following hematolymphoid malignancies or syndromes in whom allogeneic hematopoietic stem cell transplant (HST) is warranted. Specific disease categories include:

  * Indolent advanced stage non-Hodgkin lymphomas
  * Mantle cell lymphoma
  * Chronic lymphocytic leukemia
  * Hodgkin disease (Hodgkin's lymphoma)
  * Acute leukemias in complete remission
  * Aplastic anemia
  * Paroxysmal nocturnal hemoglobinuria
  * Myelodysplastic or myeloproliferative syndromes.
  * Other selected malignancies/disorders may also be considered but must be approved by the transplant team and the Principal Investigator.
* Age > 50 years, or if < 50 years of age, considered to be at high risk for regimen-related toxicity associated with conventional myeloablative transplants due to pre-existing medical conditions or prior therapy.
* A fully human leukocyte antigen (HLA)-identical sibling or matched unrelated donor is available. Potential participants with one antigen mismatched donors can be considered but only after discussion with the transplant team and the Principal Investigator.
* Participant must be competent to give consent.

EXCLUSION CRITERIA:

* Progressive hematolymphoid malignancies despite conventional therapies, or acute leukemias not in complete remission.
* Uncontrolled central nervous system (CNS) involvement with disease
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Pregnant
* Cardiac ejection fraction < 30%
* Uncontrolled cardiac failure
* Pulmonary diffusing capacity (DLCO) < 40% predicted
* Elevation of bilirubin to > 3 mg/dL
* Transaminases > 4 x the upper limit of normal
* Creatinine clearance < 50 cc/min (24-hour urine collection)
* Karnofsky performance score < 60%
* Poorly controlled hypertension on multiple antihypertensives
* Documented fungal disease that is progressive despite treatment
* HIV-positive. Other viral infections, ie, Hepatitis B- and C- positive, evaluated on a case-by-case basis
* Psychiatric disorders or psychosocial problems which in the opinion of the primary physician or Principal Investigator would place the patient at unacceptable risk from this regimen.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2003-03; Primary Completion 2014-04 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lowsky R, Takahashi T, Liu YP, Dejbakhsh-Jones S, Grumet FC, Shizuru JA, Laport GG, Stockerl-Goldstein KE, Johnston LJ, Hoppe RT, Bloch DA, Blume KG, Negrin RS, Strober S. Protective conditioning for acute graft-versus-host disease. N Engl J Med. 2005 Sep 29;353(13):1321-31. doi: 10.1056/NEJMoa050642. PMID 16192477
- [Result] Jones CD, Arai S, Lowsky R, Tyan DB, Zehnder JL, Miklos DB. Complete donor T-cell engraftment 30 days after allogeneic transplantation predicts molecular remission in high-risk chronic lymphocytic leukaemia. Br J Haematol. 2010 Sep;150(5):637-9. doi: 10.1111/j.1365-2141.2010.08252.x. Epub 2010 Jun 7. No abstract available. PMID 20528878
- [Result] Rezvani AR, Kanate AS, Efron B, Chhabra S, Kohrt HE, Shizuru JA, Laport GG, Miklos DB, Benjamin JE, Johnston LJ, Arai S, Weng WK, Negrin RS, Strober S, Lowsky R. Allogeneic hematopoietic cell transplantation after failed autologous transplant for lymphoma using TLI and anti-thymocyte globulin conditioning. Bone Marrow Transplant. 2015 Oct;50(10):1286-92. doi: 10.1038/bmt.2015.149. Epub 2015 Jul 6. PMID 26146806
- [Result] Kohrt HE, Turnbull BB, Heydari K, Shizuru JA, Laport GG, Miklos DB, Johnston LJ, Arai S, Weng WK, Hoppe RT, Lavori PW, Blume KG, Negrin RS, Strober S, Lowsky R. TLI and ATG conditioning with low risk of graft-versus-host disease retains antitumor reactions after allogeneic hematopoietic cell transplantation from related and unrelated donors. Blood. 2009 Jul 30;114(5):1099-109. doi: 10.1182/blood-2009-03-211441. Epub 2009 May 7. PMID 19423725
- [Result] Benjamin J, Chhabra S, Kohrt HE, Lavori P, Laport GG, Arai S, Johnston L, Miklos DB, Shizuru JA, Weng WK, Negrin RS, Lowsky R. Total lymphoid irradiation-antithymocyte globulin conditioning and allogeneic transplantation for patients with myelodysplastic syndromes and myeloproliferative neoplasms. Biol Blood Marrow Transplant. 2014 Jun;20(6):837-43. doi: 10.1016/j.bbmt.2014.02.023. Epub 2014 Mar 7. PMID 24607552

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-myeloablative Transplantation
Started | 303
Transplanted | 296
90 Days Post-transplant | 161
Completed | 158
Not Completed | 145
Not completed — Not Eligible | 4
Not completed — Withdrawal by Subject | 3
Not completed — Death | 138

BASELINE CHARACTERISTICS:
Arm/Group | Non-myeloablative Transplantation
Number analyzed (Participants) | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 260
  >=65 years | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 276
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 37
  Native Hawaiian or Other Pacific Islander | 7
  Black or African American | 6
  White | 233
  More than one race | 0
  Unknown or Not Reported | 20
Histology [Number; unit: participants]
  Acute Biphenotypic Leukemia | 1
  Acute Leukemia, Nos | 1
  Acute Monocytic Leukemia | 2
  Acute Myeloid Leukemia | 84
  Acute Promyelocytic Leukemia | 4
  Angioimmunoblastic T-Cell Lymphoma | 1
  B lymphoblastic leukemia/lymphoma, NOS | 1
  B-Cell Chr. Lymph. Leuk./Small Lymph. Lymphoma | 45
  Chronic Myelogenous Leukemia, Bcr/Abl Positive | 1
  Chronic Myeloid Leukemia, Nos | 8
  Chronic Myeloproliferative Disease, Nos | 2
  Cutaneous T-Cell Lymphoma, Nos | 1
  Follicular Lymphoma, Grade 1-3 | 4
  Hodgkin Lymphoma, Nodular Sclerosis, Nos | 4
  Hodgkin Lymphoma, Nos | 20
  Malignant Lymphoma, Non-Hodgkin | 86
  Mantle Cell Lymphoma | 10
  Marginal Zone B-Cell Lymphoma, Nos | 2
  Mature T-Cell Lymphoma, Nos | 1
  Ml, Large B-Cell, Diffuse | 2
  Ml, Small B Lymphocytic, Nos | 1
  Myelodysplastic Syndrome, Nos | 3
  Precursor Cell Lymphoblastic Leukemia, Nos | 15
  Prolymphocytic Leukemia, Nos | 1
  Prolymphocytic Leukemia, T-Cell Type | 1
  Subcutaneous Panniculitis-Like T-Cell Lymphoma | 1
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Acute Graft vs Host Disease (GvHD)
Description: The incidence of acute GvHD after transplantation was assessed per Glucksberg GvHD grade, a compound scale based on the following combinations of disease stages.
  Skin Stages
  * 0: No rash
  * 1: Maculopapular (MP) rash <25% of body surface area
  * 2: MP rash on 25-50% of body surface area
  * 3: Generalized erythroderma (ED)
  * 4: Generalized ED with bullous formation and desquamation
  Liver Stages (Bilirubin in mg/dL)
  * 0: <2
  * 1: 2-3
  * 2: 3.01-6
  * 3: 6.01-15.0
  * 4: >15
  Gastrointestinal (GI) Stages (diarrhea)
  * 0: None or < 500 mL/day
  * 1: 500-999 mL/day
  * 2: 1000-1499 mL/day
  * 3: >1500 mL/day
  * 4: Severe abdominal pain, with or without ileus
  Glucksberg Overall grade
  * Grade 1: Skin 1/2; GI 0; Liver 0; Karnofsky performance scale (KPS) 90-100%
  * Grade 2: Skin 1-3; GI 1; Liver 1; KPS 70-80
  * Grade 2: Skin 2/3; GI 2/3; Liver 2-4; KPS 50-60
  * Grade 4: Skin 2-4; GI 2-4; Liver 2-4; KPS 30-40
Time Frame: 100 days post-transplant
Population: Reports the incidence of Grades 2 to 4 acute GvHD, as observed for the initial 37 participants treated on this study, who constitute the Primary Analysis for the study. See linked citation Lowsky, et al. NEJM. 29Sep2005;353(13)1321-1331.
Measure: Number; unit: percentage of participants
Arm/Group | Non-myeloablative Transplantation
Number analyzed (Participants) | 37
percentage of participants | 2.7

2. Secondary Outcome: Acute Graft vs Host Disease (GvHD), All Evaluable
Description: as for outcome 1
Time Frame: 100 days post-transplant
Population: Reports data for all evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | Non-myeloablative Transplantation
Number analyzed (Participants) | 303
percentage of participants | 11

3. Secondary Outcome: Incidence of Relapse
Description: Reports the overall rate of disease relapse, occurring any time within 3 years after transplant
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Non-myeloablative Transplantation
Number analyzed (Participants) | 303
percentage of participants | 53

4. Secondary Outcome: Overall Survival (OS)
Time Frame: 3 and 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Non-myeloablative Transplantation
Number analyzed (Participants) | 303
percentage of participants
  3 years | 70
  5 years | 64

5. Secondary Outcome: Event-free Survival (EFS)
Description: Reports the number and proportion of participants who neither died due to any cause nor experienced relapse.
Time Frame: 3 and 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Non-myeloablative Transplantation
Number analyzed (Participants) | 303
Participants
  3 years | 44
  5 years | 38

6. Secondary Outcome: Transplant-related Mortality
Description: Reports the proportion of participants who expired within 1 year due to any complication or failure of the transplant.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Non-myeloablative Transplantation
Number analyzed (Participants) | 303
percentage of participants | 6

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse events other than death, secondary malignancy, or relapse were not collected.
Arm/Group | Non-myeloablative Transplantation
All-Cause Mortality (participants affected / at risk) | 138/303
Serious Adverse Events (participants affected / at risk) | 138/303
Other Adverse Events (participants affected / at risk) | 55/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-myeloablative Transplantation (N=303)
Deaths (Gastrointestinal disorders) | 138
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-myeloablative Transplantation (N=303)
Secondary malignancy (Gastrointestinal disorders) | 4 (4)
Secondary malignancy (Skin and subcutaneous tissue disorders) | 26 (26)
Secondary malignancy (Reproductive system and breast disorders) | 2 (2)
Secondary malignancy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Secondary malignancy (Blood and lymphatic system disorders) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No